CLINICAL TRIAL: NCT06320769
Title: Role of Rotational Guided Growth in Management of Increased Femoral Anteversion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24101994
Record Dates: First submitted 2024-02-23; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Increased Femoral Anteversion
Keywords: Rotational Guided Growth; Torsional Deformities; Guided Growth; Rotational Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rotational Guided Growth (Experimental): o On a radiolucent operating table with the child supine, a torniquet is applied. The limb is prepped and draped.
  oA Kirschner wire is inserted in midsagittal plane of the distal femoral physis from medial to lateral under fluoroscopic guidance.
  After the initial step, One of three Surgical techniques might be used according to surgeon preference and patient age:
  * Plate technique
  * Non-absorbable suture technique
  * Cerclage wire technique
  Interventions: Device: Plate Technique

INTERVENTIONS:
Device: Plate Technique — Using Plates, non-absorbable sutures or cerclage wires to guide the distal femoral physis towards rotational growth to correct deformity
  Other Names: Non-absorbable Suture Technique; Cerclage Wire Technique

SUMMARY:
Efficacy of guided growth in coronal plane deformity correction and limb length discrepancy has been well-established. Recently, studies have explored the validity of guided growth in correction of rotational deformity through a modified method of application.

This concept has been validated in animal studies, biomechanical studies and two limited human case series through different methods.

This study evaluates the efficacy of rotational guided growth in management of increased femoral anteversion using three different constructs.

DETAILED DESCRIPTION:
The purpose of this study is:

1. Evaluate the efficacy of different constructs in correcting increased femoral anteversion clinically and radiographically.
2. Asses possible complications of this new concept including LLD, undesired coronal, sagittal plane deformity and stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Children with increased femoral anteversion causing in-toeing with decreased agility.
* Aged 8 years and above with at least two years of bone growth remaining.

Exclusion Criteria:

* Any patient who underwent previous femoral osteotomy.
* Any patient with sick physis (skeletal dysplasias, post traumatic / post infective physeal damage, active rickets).
* Cerebral Palsy (CP) patients

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Gait | 12 months
  Foot Progression Angle 5-10 degrees by clinical gait assesment

SECONDARY OUTCOMES:
Limb length discrepancy | 12 months
  Difference between length of both limbs through clinical measurement
Angular Deformities | 12 months
  CR radiographic measuement including angles such as MPTA, LDFA

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Hassan Abdelaziz, Professor, Study Chair — Ain Shams University
Locations (1):
- Faculty of Medicine, Ainshams University, Cairo, El-Waily, Egypt

IPD SHARING:
Plan to Share IPD: No